CLINICAL TRIAL: NCT07053631
Title: Investigation of a New Window Into Intracranial Pressure: Venous Occlusion Pressure of the Isolated Periorbital Vein
Acronym: VOPxICP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Katharina Wolf, Funktionsoberärztin Leiterin der Liquorzirkulations-Ambulanz Fachärztin für Neurologie, University of Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VOPxICP pilot-study
Record Dates: First submitted 2025-04-22; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Indication for CSF Dynamic Testing; Indication for CSF Infusion Test
Keywords: ICP; non-invasive ICP assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venous occlusion pressure measurements (Experimental)
  Interventions: Device: venous occlusion pressure Measurement

INTERVENTIONS:
Device: venous occlusion pressure Measurement — non-invasive venous occlusion pressure of a targeted periorbital vein is measured in parallel to clinical standard CSF dyanmic testing including standard CSF infusiontest

SUMMARY:
Elevated intracranial pressure (ICP) occurs when pressure inside the skull rises above normal levels, potentially leading to brain damage or herniation. Monitoring ICP is critical for managing conditions like brain tumors, traumatic brain injury, and stroke. Current ICP monitoring methods are invasive and carry risks, including infection and brain damage. For less severe cases, lumbar puncture is a safer, less invasive alternative. This study explores the potential of a non-invasive method, using venous pressure near the eye, to estimate ICP. The goal is to assess whether the results from this non-invasive approach are similar to the invasive lumbar CSF pressure measurements.

DETAILED DESCRIPTION:
Elevated intracranial pressure, also known as intracranial hypertension, is a clinical condition occurring when the pressure within the cranial vault rises above physiological levels, which can eventually lead to reduced cerebral perfusion, ischemia, and potentially fatal brain herniation. Measuring intracranial pressure therefore plays a crucial role in the diagnosis and management of numerous neurological or neurosurgical pathological conditions such as brain tumors, traumatic brain injury, central nervous system infections, ischemic stroke, hydrocephalus and idiopathic intracranial hypertension. The standard of care for intracranial pressure monitoring involves invasive procedures.

This study will attempt to measure intracranial pressure by using venous occlusive pressure measured by non-invasive measurements of the isolated periorbital vein. These non-invasive measurements will be performed in parallel to invasive intracranial pressure (ICP) measurements during the current standard of care diagnostic dynamic CSF testing in patients scheduled to undergo the procedure. In addition to the primary objective, this study will also explore potential relations of the venous occlusion pressure to derivatives of dynamic CSF testing.

During the routine dynamic CSF testing, patients will be lying in the recumbent lateral position throughout the test. During the routine setup and preparation time for the CSF dynamic testing, the patient will be equipped with a pneumatic mask and one cycle of 6 successive compression sonography measurements will be demonstrated once by an investigator (#1). After this, the patient is asked to rate the discomfort of the procedure.

The mask will be deflated for the standard lumbar puncture by the physician (investigator #2). After basic testing of the opening pressure and removal of cerebrospinal fluid if needed, a monitoring and infusion setup will be connected to the lumbar needle to perform the actual dynamic CSF testing monitored by investigator #2 according to clinical routines.

Intermittent non-invasive measurements of the isolated periorbital vein will be performed by investigator #1 at regular pre-defined timepoints during this procedure (20 to 30 timepoints in total per participant), without any modification of the SOP and without impact on its duration.

A venous occlusion pressure measurement cycle itself comprises 6 successive venous occlusions and lasts no more than 30 seconds. The measurement cycle will require the investigator to inflate the mask, to identify one feasible frontal vein as the target vein, and to gently press the ultrasound probe against the target vein on the forehead of the participant six times. After this, the investigator deflates the mask is deflated, saves the recording and rates the feasibility of finding the periorbital vein.

The CSF dynamic testing is performed according to the following stages after the patient is positioned, the measurement set-ups are prepared, and after successful lumbar puncture:

1. Tilt table assessment: after a baseline period to monitor a stable ICP (2-3 minutes), lumbar ICP is measured at different tilt table angles in the following sequence: 0°, -10°, 0°, +10°, +30°. Each angle is held about 3 minutes as far as possible artifact-free. In parallel, for each angle assessed, one measurement cycle of venous occlusion pressure of the periorbital vein is performed with the mask deflated followed by one with the mask inflated. Between measurement cycles, the mask is worn deflated.
2. Baseline: lumbar ICP is measured at a 0° table tilt for about 6 minutes, as far as possible artifact-free. One measurement cycle of venous occlusion pressure of the periorbital vein is performed every 2 minutes with the mask kept inflated during the 6 minutes baseline.
3. Infusion: Constant infusion is started with a predefined rate depending on the disease investigated. The test lasts about 20 to 35 minutes. Once the infusion is stopped, final lumbar ICP measurements are continued until the measured pressure normalizes or stabilizes. One measurement cycle of venous occlusion pressure of the periorbital vein is performed with the mask inflated every 3 minutes. Between measurement cycles, the mask is worn deflated.
4. (optional) Tilt table assessment: same as phase 1 - this phase is indicated according to SOP, data collection will cover this part of the test only if performed.

   * (optional) A Queckenstedt maneuver will be performed at certain timepoints during the study with measurements of the periorbital vein with the mask inflated occurring during the maneuver.

Output measurements:

Standard of care lumbar ICP measurements are made continuously throughout the cerebrospinal fluid dynamic testing and displayed on the ICM+® software with precise timestamps and event labeling to enable synchronization with the venous occlusion pressure measurements. Mean lumbar ICP value during the 1-minute window following the start of the venous occlusion pressure measurement cycle will be taken for data analysis.

Venous occlusion pressure is determined by investigator 1 on the recorded compression ultrasound video sequence as the pressure corresponding to the first moment of full occlusion of the vein. The mean venous occlusion pressure of the periorbital vein during a measurement cycle will be used and reported for data analysis.

Expected duration of each subject's participation:

The duration of the test largely depends on the patient's individual diagnosis, time needed to perform the lumbar puncture, and findings during the test. In general, the test lasts between 45 minutes and

1h30 including all preparations. The integrated measurements of the venous occlusion pressure do not prolong the standard procedure.

PROJECT OBJECTIVES The primary objective of the project is to determine if non-invasive venous occlusion pressure measurements of the isolated target periorbital vein correlate with intracranial pressure as assessed through standard invasive lumbar CSF pressure measurements.

The secondary objectives are to investigate:

1. The relation of the venous occlusion pressure to further derivatives of the dynamic CSF testing
2. The diagnostic potential of the non-invasive method for ICP determination
3. The stability of the venous occlusion pressure of the target vein when isolated from communicating facial veins by the inflated mask
4. The alterations of venous filling pressure (mask not inflated) induced by routine tilt-table maneuvers of the CSF dynamic testing compared to the alterations of venous occlusion pressure of the isolated vein (mask inflated)
5. The feasibility of finding and compressing the target periorbital vein for the investigators during the routine tilt-table maneuvers of the CSF dynamic testing
6. The effect of re-referencing measurements by the baseline venous filling pressure (mask not inflated, horizontal recumbent lateral patient position) on the correlation with invasive lumbar ICP and diagnostic potential of the new non-invasive method.
7. The tolerability of the mask for the participants

STUDY DESIGN This study is an exploratory, single-arm intra-participant comparative and single-center project, aiming to assess the correlation between the venous occlusion pressure of the isolated periorbital frontal vein measured with compression sonography with concomitant standard of care invasive lumbar ICP in patients with CSF disturbance scheduled for CSF dynamic testing.

* Intervention: non-invasive venous occlusion pressure of the isolated periorbital frontal vein measurements using compression sonography will be compared to invasive lumbar ICP pressures obtained from standard of care cerebrospinal fluid dynamic testing procedures at pre-defined timepoints. The influence of different cofounding factors will also be assessed.
* Subjects: 10
* Intra-participant control: lumbar ICP measured continuously during standard practice
* Blinding: the operator performing the non-invasive measurements will be blinded to the invasive measurements during the cerebrospinal dynamic testing
* Duration of the investigation: 6 months
* Expected duration per participant: duration of standard of care procedure (between 45 minutes and 1 hour 30) plus time needed for self-reporting (2-3 minutes)

STUDY POPULATION Inclusion criteria

* Medical indication to perform routine craniospinal CSF dynamic testing according to standard operative procedures
* Aged 18-95
* Willing and able to provide valid signed informed consent

Exclusion Criteria

* Patients with any known ongoing, or history of, abnormal CSF communication
* Patients with any kind of prior intervention for CSF diversion
* Patients with acute brain damage within the preceding 6 months
* Patients with transdural surgery within the preceding 6 months
* Head wounds or hematoma that could hinder access to measurement site
* Any known pathological condition linked to the orbital socket influencing venous outflow

Screening and Recruitment Screening and recruitment of study participants will take place at the University Hospital Freiburg, Department of Neurosurgery. All subjects with suspected CSF disturbances who are already scheduled for cerebrospinal fluid dynamic testing will be approached and screened upon eligibility. All eligible subjects will receive participant information. As part of the participant information, the patient will be handed the mask for demonstration purposes.

Statistical analysis plan:

The statistical software package R (Version 4.0 and eventual upgrades; R Core Team) will be used throughout statistical analyses.

Data listings will include all subjects. All data exclusions, including premature terminations, will be detailed and tabulated. All data will be summarized descriptively. Quantitative variables will be described with the number of non-missing values, mean, standard deviation (SD), median, interquartile ranges and minimum/maximum values. Qualitative variables will be described with the number and percentage with 95 Confidence interval of subjects with each qualitative characteristic.

Primary objective:

The correlation of the primary endpoints will be evaluated by the Spearman correlation (rs) and rated as moderate and superior at > 0.6 and as very strong at >0.8 [33]. Additionally, a scatter plot will be provided to demonstrate the relation of the two measurements.

Furthermore, all correlations will be investigated corrected for multiple measurements applying the repeated measures correlation method (rmcorr) determining the common within-individual association for paired measures assessed on multiple timepoints across multiple individuals [34]. The correlation coefficient (rm) will be rated using the same criteria as for the spearman correlation [33].

Secondary objectives:

1. To explore potential relations of the venous occlusion pressure to derivatives of dynamic CSF testing, the following approaches will be chosen:

   * Correlation between occlusion pressure in mmHg with diastolic ICP and systolic ICP will be rated by spearman correlation. Correlation coefficients superior to 0.6 will be rated as moderate and superior to 0.8 as very strong [33].
   * A multivariable linear regression for venous occlusion testing will be constructed using the parameters derived of the CSF dynamic testing (Amplitude, Elastance, RCSF) with some evidence for a difference (p<0.2). Adjusted R-squares, Beta-coefficients with 95% CI, standard errors will be reported.
2. To assess the diagnostic potential of the new non-invasive method for ICP monitoring, the agreement between paired measurements will be evaluated using Bland Altman plots. Limits of agreement (mean difference ± 1.96 standard deviations) will be calculated, and the bias (mean difference) will be reported. Diagnostic value will be assessed based on the recommendations of the Association of Advancement of Medical Instrumentation [35]:

   * when ICP ranges between 0-20 mmHg, an absolute difference of 2mmHg is acceptable
   * when ICP is between 20 -100 mmHg, the relative difference should not exceed 10%.
3. The stability of target vein isolation from communicating veins will be assessed descriptively with the mean, standard deviation and rate of pressure drop (the difference of last and first measurement timepoint) of the repeated consecutive venous pressure measurements of the isolated periorbital vein (mask inflated) during the 6-minutes standard baseline procedure (stable invasive lumbar ICP) and by computing the intra-class correlation coefficient, two-way, mixed models.
4. To compare the alterations of the venous filling status (mask not inflated) of the participant with the venous occlusion pressure measurements of the isolated vein (mask inflated) during the standard tilt-table procedure, the difference between the mean venous occlusion pressure with the mask inflated and associated mean venous occlusion pressure measured without mask inflation will be computed for head down tilt (-10°), flat (0°) and head up tilts (+10 and +30°) and reported descriptively for each angle as median and interquartile range across participants.
5. To assess the effect of using baseline venous filling pressure (mask not inflated, 0° standard patient position) as a correction factor on the correlation and diagnostic potential of the new non-invasive method:

   The venous filling correction factor, defined as the mean venous pressure without mask inflation at 0° tilt, is subtracted from the from the pressure readings with the mask inflated The "corrected" pressure readings are used to re-compute the correlation metrics of the first endpoint and the agreement between paired measurements The "corrected" results will be compared against previous results (magnitude and fisher score for the correlation; paired t-test, pitman's test for variance and diagnostic potential criteria assessment[35] for the agreement)
6. To assess the feasibility of finding the target periorbital vein during the tilt table procedure, the investigator-reported scores for each assessed angle and participant will be described descriptively with the mean, standard deviation (SD), median, interquartile range and minimum/maximum values.
7. To assess the tolerability of the mask, participant-reported discomfort scale will be reported descriptively with the mean, standard deviation (SD), median, interquartile range and minimum/maximum values and the number/percentage of subjects with each qualitative characteristic.

ELIGIBILITY:
Inclusion Criteria:

* Medical indication to perform routine craniospinal CSF dynamic testing according to standard operative procedures
* Aged 18-95
* Willing and able to provide valid signed informed consent

Exclusion Criteria:

* Patients with any known ongoing, or history of, abnormal CSF communication
* Patients with any kind of prior intervention for CSF diversion
* Patients with acute brain damage within the preceding 6 months
* Patients with transdural surgery within the preceding 6 months
* Head wounds or hematoma that could hinder access to measurement site
* Any known pathological condition linked to the orbital socket influencing venous outflow

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Venous occlusion pressure measurement (mmHg) | 60 minutes
  Mean venous occlusion pressure of one isolated target periorbital frontal vein of 6 consecutive measurements in mmHg (mask inflated) during routine infusion test in recumbent lateral position
intracranial Pressure (ICP) in mmHg | 60 minutes
  Invasive lumbar intracranial pressure measurements in mmHg (mean over a 1-minute window aligned with start of venous occlusion measurements, in mmHg) during routine infusion test in recumbent lateral position

SECONDARY OUTCOMES:
Measurement of venous occlusive pressure in mmHg | 60 minutes
  Measurement of venous occlusive pressure in mmHg at the predefined time-points throughout the dynamic CSF test.
Measurement of average systolic ICP in mmHg | 60 minutes
  Measurement of average systolic ICP in mmHg at the predefined time-points throughout the dynamic CSF test.
Measurement of average diastolic ICP in mmHg | 60 minutes
  Measurement of average diastolic ICP in mmHg at the predefined time-points throughout the dynamic CSF test.
Relationship of venous occlusion pressure measured in mmHg compared to average ICP-Amplitude in mmHg | 60 minutes
  Relationship of venous occlusion pressure measured in mmHg compared to average ICP-Amplitude in mmHg at the predefined time-points throughout the invasive CSF infusion test.
Measurement of elastance of the craniospinal system measured in ml | 60 minutes
  Measurement of elastance of the craniospinal system in ml at the predefined time-points throughout the dynamic CSF test.
Measurement of pressure-Volume-Index in ml | 60 minutes
  Measurement of pressure-Volume-Index in ml at the predefined time-points throughout the dynamic CSF test.
Measurement of CSF outflow resistance (Rcsf) in mmHg*min/m | 60 minutes
  Measurement of CSF outflow resistance (Rcsf) in mmHg*min/m at the predefined time-points throughout the dynamic CSF test.
Measurement of pulse frequency in x/min | 60 minutes
  Measurement of pulse frequency in x/min at the predefined time-points throughout the dynamic CSF test.
Measurement of respiration frequency in x/min | 60 minutes
  Measurement of respiration frequency in x/min at the predefined time-points throughout the dynamic CSF test.
The diagnostic potential of the non-invasive method for ICP determination | 60 minutes
  Assessing the diagnostic potential of non-inasive ICP values measured by venous occlusion pressure measurement compared to the invasive ICP measurement via lumbar puncture. All measurements recorded in mmHg.
Stability of venous occlusion pressure within target vein when isolated. | 60 minutes
  Venous occlusion pressure of one isolated target periorbital frontal vein over 6 consecutive measurements with mask inflated in mmHg .
Venous filling pressure with mask inflated compared to mask not inflated. | 60 minutes
  The alterations of venous filling pressure (mask not inflated) induced by routine tilt-table maneuvers of the CSF dynamic testing compared to the alterations of venous occlusion pressure of the isolated vein (mask inflated). Measured in mmHg.
Feasability of finding and compressing the target periorbital vein for the investigators | 60 minutes
  The feasibility of finding and compressing the target periorbital vein for the investigators during the routine tilt-table maneuvers of the CSF dynamic testing. Evaluated via investigator questionnaire.
The effect of re-referencing measurements by the baseline venous filling pressure (mask not inflated, horizontal recumbent lateral patient position) correlated to invasive lumbar ICP measurements | 60 minutes
  The effect of re-referencing measurements by the baseline venous filling pressure (mask not inflated, horizontal recumbent lateral patient position) on the correlation with invasive lumbar ICP and diagnostic potential of the new non-invasive method.
The tolerability of the mask for the participants | 60 minutes
  patient feedback on the mask as based on a patient survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Neurochirurgie, Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No